CLINICAL TRIAL: NCT03434704
Title: A Phase II Trial of Allogeneic Peripheral Blood Stem Cell Transplantation From Family Haploidentical Donors in Patients With Myelodysplastic Syndrome and Acute Leukemia Under Primary Antifungal Prophylaxis With Posaconazole.
Brief Title: Peripheral Blood Stem Cell Transplantation From Family Haploidentical Donors in Patients With Myelodysplastic Syndrome and Acute Leukemia Under Primary Prophylaxis With Posaconazole
Acronym: SIR-POSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ciceri Fabio (Other)
Responsible Party: Sponsor-Investigator, Ciceri Fabio, MD, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-004423-78
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Transplant-Related Hematologic Malignancy; Leukemia, Acute; Myelodysplastic Syndromes; Graft Vs Host Disease; Fungal Infection
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Graft vs Host Disease; Mycoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Treatment (Experimental): Conditioning treatment "Thiotepa-Treosulfan-Fludarabine"; PBSC graft; GvHD prophylaxis; Primary antifungal prophylaxis.
  Interventions: Drug: Conditioning treatment "Thiotepa-Treosulfan-Fludarabine"; Procedure: PBSC graft; Drug: GvHD prophylaxis; Drug: Primary antifungal prophylaxis

INTERVENTIONS:
Drug: Conditioning treatment "Thiotepa-Treosulfan-Fludarabine" — Thiotepa iv 5 mg/kg/bid (total dose TD 10 mg/kg) day -3,-2; Treosulfan iv 14g/mq/day (TD 42 g/mq) as a single daily dose day -6, -5, -4; Fludarabine iv 30 mg/m2 (TD 150 mg/m2) day -6, -5, -4, -3, -2. Thiotepa TD 5 mg/kg and treosulfan TD 36 g/mq dose reduction according to age > 65 years.
  Other Names: TTF
Procedure: PBSC graft — (target 4-8 × 106 CD34+ cells/kg patient body weight)
Drug: GvHD prophylaxis — Sirolimus orally, monitored two times a week to maintain a target therapeutic plasma level of 8-15 ng/ml from day +5.
  Mycophenolate 15 mg/kg bid i.v. or per os day +5 through +28. Cyclophosphamide 50 mg/kg i.v. day +3+4. Mesna: >80% of the cyclophosphamide dose in 3 divided doses from day +3 daily through day +5.
Drug: Primary antifungal prophylaxis — Posaconazole delayed-release tablet [available in 100 mg tablets]: 300 mg twice daily on the first day followed by a maintenance dose of 300 mg once a day, starting on the day 0 to day 85.

SUMMARY:
SIR-POSA is a phase II trial of peripheral blood stem cell (PBSC) transplantation from a partially compatible family (Haplo) donor in patients with a blood tumor (myelodysplastic syndrome (MDS) and acute leukemia) treated for the prevention of primary fungal infections with posaconazole.

The aim is evaluate the composite end-point graft-versus-host disease-free, relapse-free survival (GRFS) in these patients and evaluate the feasibility and efficacy of posaconazole oral tablets as primary antifungal prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of myelodysplastic syndromes or acute leukemia
* Activation of an alternative donor search by the Italian Bone Marrow Donor Registry (IBMDR) with absence of a 10/10 Human Leukocyte Antigens (HLA) matched unrelated donor
* Age >18
* Unavailability of a HLA-matched related donor (MRD)
* Performance status : Eastern Cooperative Oncology Group (ECOG) <3
* Written and signed informed consent
* Life expectancy not severely limited by concomitant illness.

Exclusion Criteria:

* Women of child-bearing potential who do not agree to abstinence or, if sexually active, do not agree to the use of highly effective method of birth control such as condoms, implants, injectables, combined oral contraceptives, intrauterine devices (IUDs), vasectomised partner on treatment and for at least 6 months thereafter.
* Pregnant or nursing (lactating) women.
* Known allergies, hypersensitivity, or intolerance to any experimental drugs.
* Any active, uncontrolled infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-10-13 (Actual); Study Completion 2019-10-13 (Actual)

PRIMARY OUTCOMES:
Graft-versus-host disease-free, relapse-free survival (GRFS) | 2 years
  GRFS events is defined as the first event among grade III-IV acute Graft vs. Host Disease (GVHD), severe chronic GVHD, relapse and death from any cause

SECONDARY OUTCOMES:
Efficacy of antifungal prophylaxis strategy | 85 days after transplantation
  The rate of proven, probable and possible invasive fungal diseases documented within the first 85 days after transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele, Milan, Lombardy, Italy